CLINICAL TRIAL: NCT01623921
Title: Statins and Selective Cyclooxygenase-2 Receptor Inhibitors in Blunt Chest Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Director, Division of Research & Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-08-WAA-026911-TLV
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Blunt Chest Trauma; Acute Respiratory Distress Syndrome
Keywords: Lung; Contusion; Injury; Cyclooxygenase; Statin
MeSH Terms: conditions — Respiratory Distress Syndrome; Contusions; Wounds and Injuries | interventions — Celecoxib; Rosuvastatin Calcium; Psychotherapy, Multiple

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- control (Other): Group 1: control :(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Interventions: Drug: standard care treatment
- Celecoxib (Active Comparator): Group 2: Celecoxib 200 mg × 2/d+:(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Interventions: Drug: Celecoxib
- rosuvastatin (Active Comparator): Group 3: Rosuvastatin 40mg × 1/d+:(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Interventions: Drug: Rosuvastatin
- Combined therapy (Active Comparator): Group 4: Combined therapy with Celecoxib 200 mg× 2/d + Rosuvastatin 40× 1/d +:(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Interventions: Drug: Combined therapy

INTERVENTIONS:
Drug: standard care treatment — Group 1: control :(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Arms: control
Drug: Celecoxib — Celecoxib 200 mg × 2/d+:(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Arms: Celecoxib
Drug: Rosuvastatin — Rosuvastatin 40mg × 1/d+:(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Arms: rosuvastatin
Drug: Combined therapy — Combined therapy with Celecoxib 200 mg× 2/d + Rosuvastatin 40× 1/d +:(standard care treatment for individual lung contusion inluding analgesia with paracetamol/dypiron/ tramal)
  Arms: Combined therapy

SUMMARY:
Background: Lung contusion affects 17%-25% of adult blunt trauma patients, and is the leading cause of death from blunt thoracic injury. Statins are lipid-lowering drugs with recently suggested anti-inflammatory and antioxidant properties. Cyclo-oxygenase-2 (COX-2) is a key enzyme in the production of prostaglandins (PG), and evidence suggests that COX-2 plays an important role in the pathogenesis of acute lung injury (ALI).

Aims: The current study aims at evaluating the beneficial effects of statins and COX-2 receptor inhibitors on ALI elicited by blunt trauma to the chest.

Methods: After approval by the institutional ethics and a scientific committee, and obtaining informed consent , patients admitted to the emergency department (ED) due to blunt trauma with a diagnosis of lung contusion will be enrolled in the study.The effects of statins and COX 2 inhibitors on ALI will be assessed by recording clinical parameters and measuring inflammatory mediators levels in the serum and in the bronchoalveolar space.

Expected results: The investigators expect to find that the proposed treatment will be effective in reducing ALI burden. The investigators also suppose that using a combination of those drugs will synergistically potentiate their effect on ALI.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Diagnosis of lung contusion by physical examination, chest xrays, history by the patient, accompanying persons or police.
* Ability to understand and accept the trial procedures and to sign an informed consent form in accordance with national legislation.
* Admission to ward

Exclusion Criteria:

* Penetrating trauma
* Current use of lipid-lowering therapy, use of non steroidal anti-inflammatory drugs.
* Current use of postmenopausal hormone-replacement therapy
* Evidence of hepatic dysfunction (an alanine aminotransferase level more than twice the upper limit of the normal range), a creatine kinase level more than three times the upper limit of the normal range.
* Creatinine level higher than 2.0 mg/dl
* Known uncontrolled hypertension (systolic blood pressure >190 mm Hg or diastolic blood pressure >100 mm Hg
* History of uncontrolled hypothyroidism (thyroid-stimulating hormone level> 1.5 times the upper limit of the normal range)
* Psychiatric disorders
* Pregnancy
* Known allergy or intolerance to one of the protocol drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
1. Signs of ALI, i.e., pneumonia, adult respiratory distress syndrome [ARDS] | 3 days
  1. Signs of ALI, i.e., pneumonia, adult respiratory distress syndrome [ARDS] according to following criteria:
  1. Suspected or proven infection
  2. Hypoxemia: PaO2/FiO2is ≤300 mm HgBilateral infiltrates consistent with pulmonary edema
  3. Positive-pressure mechanical ventilation through an endotracheal tube
  4. No clinical evidence of left atrial hypertension to explain bilateral infiltrates
  5. Presence of at least three of the four SIRS criteria. If only two criteria are evidenced, one must be temperature or WBC

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel